CLINICAL TRIAL: NCT07178899
Title: Designing a Smoking Intervention for Youth Smokers Using Q-Methodology: A Pilot Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHEUNG, Cara Hor Yine, Post Doctoral Fellow, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08230208
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Smoking (Tobacco) Addiction; Young Adult; RCT
Keywords: Smoking Cessation; Young Adult; RCT
MeSH Terms: conditions — Smoking; Behavior, Addictive; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: two arms: intervention group & control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the intervention group, in addition to routine counselling (15-30 minutes), they will classify their identity with our screening tool (developed in Phase 2) and then apply the counselling protocol for the participants (5-10 minutes). After the counselling session, the personalized e-messages will be sent to the participants by the counsellor for 4 weeks.
  Interventions: Behavioral: typology-based intervention
- Control Group (Active Comparator): In the control group, the routine smoking cessation counselling, including generic advice on preventing smoking relapse, will be retained, and they will receive brief e-messages that only consist of general quit advice for 4 weeks.
  Interventions: Behavioral: Routine Treatment

INTERVENTIONS:
Behavioral: typology-based intervention — The typology-based intervention includes: (1) typology-based counselling, (2) personalized E-message based on the counselling content discussed (3) a booklet introducing the typology of quit identity. All interventions and materials are delivered by smoking counselling.
  Arms: Intervention group
Behavioral: Routine Treatment — The routine smoking cessation intervention includes: (1) Routine counselling generic advice on preventing smoking relapse (2) Brief e-messages that consist of general quit advice for 4 weeks. Counsellors implement both routine practices.
  Arms: Control Group

SUMMARY:
This study aims to develop a typology-based intervention delivered by smoking cessation (SC) counsellors to prevent smoking relapse in ex-smokers who recently quit. The two main research questions include (1) Can a typology-based smoking relapse prevention intervention be feasible and accepted by the smokers and SC counsellors who deliver the new intervention? (2) What is the preliminary evidence on the efficacy of the typology-based smoking relapse prevention to increase tobacco abstinence in ex-smokers who have recently quit? If the intervention shows at least a small effect size (i.e. risk ratio>1.3), or the intervention is feasible while modifications can potentially increase the efficacy, a future definitive RCT is warranted.

DETAILED DESCRIPTION:
Phase 1 Q-method outcomes The outcomes of Phase 1 of this study will be Q-sorts completed by participants which will be inter-correlated producing a matrix for factor rotation and automatic flagging, and the z-score and the factor of the Q-sorts will be calculated.

The tobacco epidemic remains a pressing global health challenge, with tobacco-related illness contributing significantly to a high death rate worldwide. Smoking is the predominant mode of tobacco consumption worldwide and serves as the driving force behind this epidemic. According to the World Health Organization [1], there are an estimated 1.3 billion tobacco users worldwide currently. In Hong Kong, the smoking rate is estimated to be around 9.5%, with approximately 580 000 daily smokers in 2021 [2]. Despite the rate has decreased significantly from 23.3% in 1982, the Hong Kong government aims to further reduce the prevalence from 9.5% to 7.8% in 2025. The high prevalence of smoking imposes a significant public health burden worldwide, with tobacco use killing up to 50% of its users [3]. Additionally, smoking causes cancers, stroke, cardiovascular diseases and respiratory diseases [4], with around 7000 deaths reported each year [5]. One approach to reduce the smoking prevalence is to promote smoking cessation (SC) treatment among current smokers.

Young smokers constitute a large cohort of new smokers every year. It is estimated that up to 90% of daily smokers first tried smoking before 18 years old [6]. Published studies consistently highlight the concerning prevalence of youth smoking within our community. Data from the recent school survey [7] highlighted that despite only 1.2% of secondary school engages in smoking, a significant portion (7.4%, equivalent to around 24 000 students) of the youth population have previously engaged in smoking behaviour. The rate of youth ever smokers remain high at 7.4% in Hong Kong [2], equivalent to approximately 24 000 secondary school students, suggesting that youths are eagerly experimenting. This is also evident in the high prevalence of youths trying other tobacco products such as e-cigarettes or heated tobacco products, from 57.4% (178/310) in 2017 to 2018 to 85.9% (243/283) in 2019 to 2020 [8]. The shift from occasional smoking to dependency in youth is a crucial stage, making the adolescent years a key period for understanding and addressing smoking behaviours. It represents a key window for targeted interventions to prevent the progression towards regular smoking habits.

Smoking imposes severe health risks and long-term consequences. Effects of tobacco are well demonstrated [9] including the effects of nicotine on brain development [10]. The prevalence of tobacco use among youths not only jeopardizes their immediate health but negatively impacts their future well-being [11]. Moreover, observations from our communities [12] further emphasize the pressing need for effective SC initiatives tailored to the unique needs of youths. The multifaceted challenges such as peer pressure and social influences are faced by struggling youths.

In response to these identified needs, it is imperative to develop comprehensive youth-orientated SC programs that encompass various aspects of prevention, intervention and support. Evidence-based strategies such as counselling services [13] have shown promising outcomes in promoting smoke-free lifestyles among youths. Additionally, collaborations among healthcare institutions, government agencies and community organizations are crucial for maximizing the reach and effectiveness of cessation efforts. By addressing the health needs of our local community through targeted youth SC initiatives, we can significantly mitigate the adverse health effects of tobacco use among our young population.

Phase 3 Randomized control trial outcomes The primary outcomes of Phase 3 of this study will be smokers' (1) self-reported abstinence in the past 30 days at 2-month follow-up; (2) iScreen OFD Cotinine Saliva Test Kit (<30ng/ml) biochemical validated tobacco abstinence; (3) the difference of the feasibility and acceptability score of the typology-based intervention between the intervention and control group.

ELIGIBILITY:
Inclusion Criteria (Phase 1):

* Hong Kong citizens
* Have ever habitually used conventional cigarettes in the past year
* Not using cigarettes for the past 7 days
* Aged 18-25
* No barriers in communicating in Cantonese and reading and writing Chinese
* Quit smoking without using cessation services

Inclusion Criteria (Phase 3):

* Hong Kong citizens
* Have ever habitually used conventional cigarettes in the past year
* Received at least 4 weeks of smoking cessation service before enrolling into the study
* abstained from tobacco use for 7 to 30 days without using any cessation services
* Aged 18-25
* No barriers in communicating in Cantonese and reading and writing Chinese

Exclusion Criteria (Phase 1 & 3):

* Have unstable physical or psychological conditions as advised by doctors or counsellors
* Are users of illicit drugs (e.g., heroin, marijuana, ketamine, etc.)
* Have become pregnant in the past two months
* unable to communicate in Cantonese and read Chinese

Inclusion Criteria (Phase 2) (for SC counsellors) :

* SC counsellors from local SC clinics under HKU Youth Quit Line, Tung Wah Group of Hospitals Integrated Center on Smoking Cessation and United Christian Nethersole Community Health Service

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
self-reported abstinence in the past 30 days at 2-month follow-up | 2 mouths
iScreen OFD Cotinine Saliva Test Kit (<30ng/ml) biochemical validated tobacco abstinence | 2 months
  Participants who report tobacco abstinence will be invited for a biochemical validation to test if his/her saliva cotinine is less than 30ng/ml measured by the iScreen OFD Cotinine Saliva Test Kit.
the difference of the feasibility and acceptability score of the typology-based intervention between the intervention and control group. | 2 months
  We will have 4 feasibility questions and 4 appropriateness questions for counsellor to answer from 1 (Completely disagree) to 5 (Completely agree). Also, we will have 4 acceptability questions for ex-smokers to answer. We would like to observe if there is a difference between the intervention group and the control group

SECONDARY OUTCOMES:
Time required for the counselling | End of all follow-up (approximately 6 month)
  The average time required for the typological counselling in minutes
Compliance rate of the SC counsellors in following the intervention protocol | End of all follow-up (approximately 6 month)
  There were 26 questions in the counselling protocol. SC counsellors have to record the number of questions asked during the typological counselling. The rate is calculated by "number of questions asked"/26
Proportion of screened clients who participate in the RCT | End of all follow-up (approximately 6 month)
  The proportion is calculated by "Number of enrolled participants" / "Total number of participant screened"
Dropout rate of the participants who consent to the RCT | End of all follow-up (approximately 6 month)
  The dropout rate is calculated by "Number of participants dropout from study" / "Total number of enrolled participant"
Satisfaction on the SC counsellors | 2 months
  Satisfaction on the SC counsellors is measured by a 5 point Likert scale reported by the enrolled participants.
Satisfaction on the e-messages | 2 months
  Satisfaction on the e-messages is measured by a 10 point Likert scale reported by the enrolled participants.
Frequency of reading the e-messages | 2 months
  The Frequency of reading the e-messages is measured by 5 point Likert scale, which includes the option (5) I read all of them, (4) I read most of them, (3) I read half of them, (2) I read some of them, and (1) I read none of them.
Perceived effectiveness on the intervention | 2 months
  The perceived effectiveness on the intervention is measured by a 10 point likert scale. Participant will rate the usefulness of the messages in helping them to maintain smoking abstinence (10: Very useful | 0: Useless).
Satisfaction on the enrolment procedures | 2 months
  Satisfaction on the enrolment procedures is measured by a 10 point Likert scale reported by the participants (0: The enrollment procedure is slow and complicated | 10: the enrollment procedure is fast and simple).
Intention to recommend the intervention to other smokers | 2 months
  Intention to recommend the intervention to other smokers is measured by a 10 point Likert scale, 10: strongly recommended to other smokers | 0: not recommended to other smoker
Satisfaction about the intervention from SC counsellor | End of all follow-up (approximately 6 month)
  Satisfaction about the intervention from SC counsellor is measured by a 5 point Likert scale. SC counsellor will rate the effectiveness of the typological counselling in helping their client to quit smoking, from 1: very ineffective to 5: very effective.
Perceived appropriateness of the intervention length from SC counsellor | End of all follow-up (approximately 6 month)
  The perceived appropriateness of the intervention length from SC counsellor is measured by a 5 point Likert scale. SC counsellor will be asked if they agreed that the length of the typological counselling is suitable for their client, from 1 strongly disagree to 5 strongly agree.
Satisfaction on the enrolment and counselling procedures from SC counsellors | End of all follow-up (approximately 6 month)
  The satisfaction on the enrolment procedures from SC counsellors is measured by a 5 point Likert scale. Counsellors will be asked if they agreed that enrolment and counselling procedures is simple and could be easily done in the SC clinics, from 1: strongly disagree to 5: strongly agree.
Perceived effectiveness of the screening tool from SC counsellor | End of all follow-up (approximately 6 month)
  The perceived effectiveness of the screening tool from SC counsellor is measured by a 5 point Likert scale. SC counsellor will be asked if they agreed that the typological intervention can help them screen out smokers who are prone to relapse, from 1: strongly disagree to 5: strongly agree.
Perceived clients' acceptance of the intervention from SC counsellor | 2 months
  The Perceived clients' acceptance of the intervention from SC counsellor is measured by a 5 point Likert scale. Participants are asked if they agreed that counselling content provided the SC counselling gain their trust and acceptance, from 1: strongly disagree to 5: strongly agree.
Intention to apply this intervention in other clients from SC counsellors | End of all follow-up (approximately 6 month)
  Intention to apply this intervention in other clients from SC counsellors is measured by a 5 point Likert scale. SC counsellors are asked if they want to apply the typological intervention to other clients in future, 1: I will not apply it to my client in the future, 5: I want to apply it my client in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- LKS Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years after the completion of the relevant publications

REFERENCES:
- [Background] Zabala A, Pascual U. Bootstrapping Q Methodology to Improve the Understanding of Human Perspectives. PLoS One. 2016 Feb 4;11(2):e0148087. doi: 10.1371/journal.pone.0148087. eCollection 2016. PMID 26845694
- [Background] Watts S, Stenner P. Doing the fieldwork: participants, materials and procedure. 2012 2022/03/11. In: Doing Q Methodological Research: Theory, Method and Interpretation . London: SAGE Publications Ltd
- [Background] Karpinski JP, Timpe EM, Lubsch L. Smoking cessation treatment for adolescents. J Pediatr Pharmacol Ther. 2010 Oct;15(4):249-63. PMID 22477813
- [Background] Bailey SR, Crew EE, Riske EC, Ammerman S, Robinson TN, Killen JD. Efficacy and tolerability of pharmacotherapies to aid smoking cessation in adolescents. Paediatr Drugs. 2012 Apr 1;14(2):91-108. doi: 10.2165/11594370-000000000-00000. PMID 22248234
- [Background] Duncan Millar J, Mason H, Kidd L. What is Q methodology? Evid Based Nurs. 2022 Jul;25(3):77-78. doi: 10.1136/ebnurs-2022-103568. Epub 2022 May 24. No abstract available. PMID 35609957
- [Background] Bowen NK, Lee JS, Weller BE. SOCIAL ENVIRONMENTAL RISK AND PROTECTION: A TYPOLOGY WITH IMPLICATIONS FOR PRACTICE IN ELEMENTARY SCHOOLS. Child Sch. 2007;29(4):229-242. doi: 10.1093/cs/29.4.229. PMID 21709821
- [Background] Tombor I, Shahab L, Herbec A, Neale J, Michie S, West R. Smoker identity and its potential role in young adults' smoking behavior: A meta-ethnography. Health Psychol. 2015 Oct;34(10):992-1003. doi: 10.1037/hea0000191. Epub 2015 Jan 26. PMID 25622078
- [Background] Jarvelaid M. Adolescent tobacco smoking and associated psychosocial health risk factors. Scand J Prim Health Care. 2004 Mar;22(1):50-3. doi: 10.1080/02813430310000988. PMID 15119521
- [Background] Tombor I, Vangeli E, West R, Shahab L. Progression towards smoking cessation: Qualitative analysis of successful, unsuccessful, and never quitters. J Subst Use. 2017 Oct 5;23(2):214-222. doi: 10.1080/14659891.2017.1378746. eCollection 2018. PMID 29527597
- [Background] Rose JS, Chassin L, Presson C, Sherman SJ, Stein MD, Col N. A latent class typology of young women smokers. Addiction. 2007 Aug;102(8):1310-9. doi: 10.1111/j.1360-0443.2007.01889.x. PMID 17624981
- [Background] Thomas JL, Luo X, Bengtson J, Wang Q, Ghidei W, Nyman J, Lust K, An L, Wetter DW, Epstein L, Ahluwalia JS. Enhancing Quit & Win contests to improve cessation among college smokers: a randomized clinical trial. Addiction. 2016 Feb;111(2):331-9. doi: 10.1111/add.13144. Epub 2015 Nov 11. PMID 26767340
- [Background] Villanti AC, West JC, Klemperer EM, Graham AL, Mays D, Mermelstein RJ, Higgins ST. Smoking-Cessation Interventions for U.S. Young Adults: Updated Systematic Review. Am J Prev Med. 2020 Jul;59(1):123-136. doi: 10.1016/j.amepre.2020.01.021. Epub 2020 May 14. PMID 32418800
- [Background] Chaiton M, Diemert L, Cohen JE, Bondy SJ, Selby P, Philipneri A, Schwartz R. Estimating the number of quit attempts it takes to quit smoking successfully in a longitudinal cohort of smokers. BMJ Open. 2016 Jun 9;6(6):e011045. doi: 10.1136/bmjopen-2016-011045. PMID 27288378
- [Background] Rosa JD, Aloise-Young P. A Qualitative Study of Smoker Identity Among College Student Smokers. Subst Use Misuse. 2015;50(12):1510-7. doi: 10.3109/10826084.2015.1018549. Epub 2015 Nov 19. PMID 26584272
- [Background] Davey, G. and Zhao, X. (2020), Turning Points to Becoming a Tobacco Smoker: Smoking Initiation and Identity Change among Chinese Youth. Symbolic Interaction, 43: 308-331
- [Background] Bitar S, Collonnaz M, O'Loughlin J, Kestens Y, Ricci L, Martini H, Agrinier N, Minary L. A Systematic Review of Qualitative Studies on Factors Associated With Smoking Cessation Among Adolescents and Young Adults. Nicotine Tob Res. 2024 Jan 1;26(1):2-11. doi: 10.1093/ntr/ntad167. PMID 37648287
- [Background] Barrington-Trimis JL, Braymiller JL, Unger JB, McConnell R, Stokes A, Leventhal AM, Sargent JD, Samet JM, Goodwin RD. Trends in the Age of Cigarette Smoking Initiation Among Young Adults in the US From 2002 to 2018. JAMA Netw Open. 2020 Oct 1;3(10):e2019022. doi: 10.1001/jamanetworkopen.2020.19022. PMID 33021650
- [Background] An LC, Klatt C, Perry CL, Lein EB, Hennrikus DJ, Pallonen UE, Bliss RL, Lando HA, Farley DM, Ahluwalia JS, Ehlinger EP. The RealU online cessation intervention for college smokers: a randomized controlled trial. Prev Med. 2008 Aug;47(2):194-9. doi: 10.1016/j.ypmed.2008.04.011. Epub 2008 May 2. PMID 18565577
- [Background] Cho ER, Brill IK, Gram IT, Brown PE, Jha P. Smoking Cessation and Short- and Longer-Term Mortality. NEJM Evid. 2024 Mar;3(3):EVIDoa2300272. doi: 10.1056/EVIDoa2300272. Epub 2024 Feb 8. PMID 38329816
- [Background] Li WHC, Chan SSC, Wang MP, Ho KY, Cheung YTY, Chan VWF, Lam TH. An Evaluation of the Youth Quitline Service Young Hong Kong Smokers. J Adolesc Health. 2017 May;60(5):584-591. doi: 10.1016/j.jadohealth.2016.11.022. Epub 2017 Jan 19. PMID 28111012
- [Background] Ho SY, Chen J, Leung LT, Mok HY, Wang L, Wang MP, Lam TH. Adolescent Smoking in Hong Kong: Prevalence, Psychosocial Correlates, and Prevention. J Adolesc Health. 2019 Jun;64(6S):S19-S27. doi: 10.1016/j.jadohealth.2019.01.003. PMID 31122545
- [Background] McClure LA, Arheart KL, Lee DJ, Sly DF, Dietz NA. Young adult former ever smokers: the role of type of smoker, quit attempts, quit aids, attitudes/beliefs, and demographics. Prev Med. 2013 Nov;57(5):690-5. doi: 10.1016/j.ypmed.2013.08.028. Epub 2013 Sep 8. PMID 24021991
- [Background] Goriounova NA, Mansvelder HD. Short- and long-term consequences of nicotine exposure during adolescence for prefrontal cortex neuronal network function. Cold Spring Harb Perspect Med. 2012 Dec 1;2(12):a012120. doi: 10.1101/cshperspect.a012120. PMID 22983224
- [Background] School of Public Health of the University of Hong Kong. School-based survey on smoking among students in 2020/21.
- [Background] US Department of Health and Human Services. Preventing Tobacco Use Among Youth and Young Adults: A Report of the Surgeon General. Atlanta, GA: US Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, Office on Smoking and Health; 2012.
- [Background] Rigotti NA, Kruse GR, Livingstone-Banks J, Hartmann-Boyce J. Treatment of Tobacco Smoking: A Review. JAMA. 2022 Feb 8;327(6):566-577. doi: 10.1001/jama.2022.0395. PMID 35133411
- [Background] World Health Organization. WHO Report on the Global Tobacco Epidemic, 2019: Offer help to quit tobacco use. Geneva: World Health Organization; 2019
- [Background] McGhee SM, Ho LM, Lapsley HM, Chau J, Cheung WL, Ho SY, Pow M, Lam TH, Hedley AJ. Cost of tobacco-related diseases, including passive smoking, in Hong Kong. Tob Control. 2006 Apr;15(2):125-30. doi: 10.1136/tc.2005.013292. PMID 16565461